CLINICAL TRIAL: NCT05912296
Title: A Randomized, Single Blind, Placebo Controlled, Single Center Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Pharmacodynamics of Single and Multiple Ascending Doses of Subcutaneously Administered RBD7022 in Participants With Normal or Elevated LDL-c Cholesterol
Brief Title: A Single and Multiple Ascending Doses Study to Evaluate the Safety, Tolerability and Pharmacokinetics of RBD7022
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Ribo Life Science Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: RBD7022
Record Dates: First submitted 2023-05-21; First posted 2023-06-22 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Hyperlipemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- RBD7022 SAD experimental group (Experimental): Subjects in SAD experimental groups will receive a single subcutaneous injection of RBD7022 on Day 0.
  Interventions: Drug: RBD7022
- RBD7022 MAD experimental group (Experimental): Subjects in MAD experimental groups will receive one subcutaneous injection of RBD7022 on Day 0 and another subcutaneous injection of RBD7022 on Day 28.
  Interventions: Drug: RBD7022
- Placebo SAD group (Placebo Comparator): Subjects in SAD placebo groups will receive a single subcutaneous injection of placebo on Day 0.
  Interventions: Drug: Placebo
- Placebo MAD group (Placebo Comparator): Subjects in MAD placebo groups will receive one subcutaneous injection of placebo on Day 0 and another subcutaneous injection of placebo on Day 28 .
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RBD7022 — Subcutaneously Administered RBD7022 in Healthy Subjects.
  Arms: RBD7022 SAD experimental group
Drug: RBD7022 — Subcutaneously Administered RBD7022 in Healthy Subjects.
  Arms: RBD7022 MAD experimental group
Drug: Placebo — Subcutaneously Administered Placebo in Healthys Subject.
  Arms: Placebo SAD group
Drug: Placebo — Subcutaneously Administered Placebo in Healthys Subject.
  Arms: Placebo MAD group

SUMMARY:
This is a randomized, single blind, placebo controlled, single center phase I study to evaluate the safety, tolerability, pharmacokinetics, and preliminary pharmacodynamics of single and multiple ascending doses of subcutaneously administered RBD7022 in participants with normal or elevated LDL-c cholesterol. The study will be performed in 2 phases: single ascending dose (SAD) phase and multiple ascending doses (MAD) phase in participants. The decision to escalate to subsequent dose levels will be made by the SRC based on the review of all available safety information in each cohort.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, aged 18 to 65 years, inclusive
* Body mass index between 17 and 28 kg/m2 , inclusive
* LDL-C normal or elevated at screening and baseline.
* Willing to comply with protocol required visit schedule and visit requirements and provide written informed consent.
* The clinical laboratory examination of the subjects was within the normal range, or abnormal but had no clinical significance as judged by the investigators, and did not affect the study results;
* Vital signs, physical examination, ECG, ultrasound showed normal or abnormal but no clinically significant as determined by the investigator.

Exclusion Criteria:

* With a clear history of primary diseases of major organs, the subject is not suitable to participate in this study considered by the investigator;
* Diagnosis of diabetes mellitus;
* Pregnant or breastfeeding women;
* Any conditions which, in the opinion of the Investigator, would make the subject unsuitable for enrollment or could interfere with the subject's participation in or completion of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Related Adverse Events as Assessed by CTCAE v5.0 | SAD up to Day 180; MAD up to Day 208
  By the examination of vital signs, physical examination, 12-lead electrocardiogram (ECG), and laboratory examination, the investigator will make an assessment of intensity for each AE and SAE reported during the study according to CTCAE V5.0

SECONDARY OUTCOMES:
The serum LDL-C level after subject dosing RBD7022 | SAD up to Day 180; MAD up to Day 208
  measure the LDL-C level in blood by lab examination and eveluate the effect of RBD7022 on Circulating LDL-c Levels (Determination of % Lowering of LDL-c to treatment/Baseline LDL-c Level)
The serum PCSK9 level after subject dosing RBD7022 | SAD up to Day 180; MAD up to Day 208
  measure the pcsk9 level in blood by lab examination and eveluate the effect of RBD7022 on Circulating PCSK9 Levels (Determination of % Lowering of PCSK9 to treatment/Baseline PCSK9 Level).
Other blood lipoprotein and lipid parameters besides LDL-c | SAD up to Day 180; MAD up to Day 208
  measure other blood lipoprotein and lipid parameters besides LDL-c in blood by lab examination and eveluate % change and absolute change in other lipoprotein and lipid parameters（TC、TG、Lp (a)、HDL-C、non HDL-C、Apo B、Apo A1、Apo A 1/ Apo B ratio） from baseline up to Day 208
The effect of RBD7022 monotherapy or RBD7022 combination with statin in patients with elevated LDL-C | SAD up to Day 180; MAD up to Day 208
  measure the LDL-C and pcsk9 level in blood by lab examination and assess % change and absolute change in LDL-c and PCSK9 from baseline up to Day 208
To characterize the pharmacokinetic parameter Cmax | SAD: within 60 min before dosing, and at 15min, 30min, 1, 2, 4, 6, 8,12, 24, 48 and 72 hours after dosing; MAD: within 60 minutes before day 0 and day 28 dosing, and at 15min, 30min, 1, 2, 4, 6, 8,12, 24 ,48 and 72 hours after Day 0 and day 28 dosing
  Plasma Maximum concentration (Cmax)
To characterize the pharmacokinetic parameter Tmax | SAD: within 60 min before dosing, and at 15min, 30min, 1, 2, 4, 6, 8,12, 24, 48 and 72 hours after dosing; MAD: within 60 minutes before day 0 and day 28 dosing, and at 15min, 30min, 1, 2, 4, 6, 8,12, 24 ,48 and 72 hours after Day 0 and day 28 dosing
  Time to maximum concentration (Tmax)
To characterize the pharmacokinetic parameter AUC0-t | SAD: within 60 min before dosing, and at 15min, 30min, 1, 2, 4, 6, 8,12, 24, 48 and 72 hours after dosing; MAD: within 60 minutes before day 0 and day 28 dosing, and at 15min, 30min, 1, 2, 4, 6, 8,12, 24 ,48 and 72 hours after Day 0 and day 28 dosing
  Area under the concentration-time curve from 0 to the collection time t (AUC0-t)
To characterize the pharmacokinetic parameter t1/2 | SAD: within 60 min before dosing, and at 15min, 30min, 1, 2, 4, 6, 8,12, 24, 48 and 72 hours after dosing; MAD: within 60 minutes before day 0 and day 28 dosing, and at 15min, 30min, 1, 2, 4, 6, 8,12, 24 ,48 and 72 hours after Day 0 and day 28 dosing
  Half-Life (t1/2)
To characterize the pharmacokinetic parameter λz | SAD: within 60 min before dosing, and at 15min, 30min, 1, 2, 4, 6, 8,12, 24, 48 and 72 hours after dosing; MAD: within 60 minutes before day 0 and day 28 dosing, and at 15min, 30min, 1, 2, 4, 6, 8,12, 24 ,48 and 72 hours after Day 0 and day 28 dosing
  Elimination rate constant (λz)
To characterize the pharmacokinetic parameter CL/F | SAD: within 60 min before dosing, and at 15min, 30min, 1, 2, 4, 6, 8,12, 24, 48 and 72 hours after dosing; MAD: within 60 minutes before day 0 and day 28 dosing, and at 15min, 30min, 1, 2, 4, 6, 8,12, 24 ,48 and 72 hours after Day 0 and day 28 dosing
  Oral clearance (CL/F)
To characterize the pharmacokinetic parameter Vz/F | SAD: within 60 min before dosing, and at 15min, 30min, 1, 2, 4, 6, 8,12, 24, 48 and 72 hours after dosing; MAD: within 60 minutes before day 0 and day 28 dosing, and at 15min, 30min, 1, 2, 4, 6, 8,12, 24 ,48 and 72 hours after Day 0 and day 28 dosing
  Volume of distribution in the terminal elimination period (Vz/F)
To characterize the pharmacokinetic parameter AUC0-inf | SAD: within 60 min before dosing, and at 15min, 30min, 1, 2, 4, 6, 8,12, 24, 48 and 72 hours after dosing; MAD: within 60 minutes before day 0 and day 28 dosing, and at 15min, 30min, 1, 2, 4, 6, 8,12, 24 ,48 and 72 hours after Day 0 and day 28 dosing
  Area under the concentration-time curve from 0 to infinity

CONTACTS AND LOCATIONS:
Overall Officials: Rui Chen, Doctor, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No